CLINICAL TRIAL: NCT02179853
Title: Anakinra in Infants and Children With Coronary Artery Abnormalities in Acute Kawasaki Disease
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: Boston Children's Hospital (Other); Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Adriana H. Tremoulet, Associate Professor, University of California, San Diego
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KD Anakinra
Record Dates: First submitted 2014-06-28; First posted 2014-07-02 (Estimated); Results first posted 2024-03-04 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2024-03

CONDITIONS: Kawasaki Disease
Keywords: Kawasaki disease; Anakinra; IL-1
MeSH Terms: conditions — Mucocutaneous Lymph Node Syndrome | interventions — Interleukin 1 Receptor Antagonist Protein

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Anakinra (Experimental): This is a dose escalation study (4 mg/kg, 6 mg/kg and 8 mg/kg).
  Interventions: Drug: Anakinra

INTERVENTIONS:
Drug: Anakinra — First two doses IV followed by SQ dosing
  Other Names: Kineret

SUMMARY:
Kawasaki disease (KD) is the leading cause of acquired heart disease in children in the developed world. Despite available treatment, 25% of children in San Diego County appropriately treated for KD develop coronary artery abnormalities that may lead to complications later in life, including heart attack. Although the investigators can identify children with KD that have these coronary artery abnormalities, there is no approved additional treatment to decrease coronary artery inflammation and arrest or prevent damage to the coronary arteries. Anakinra, a therapy that blocks the high levels of interleukin 1 (IL1) that lead to inflammation during acute KD, has been shown in the KD mouse model to prevent the development of coronary artery damage. Therefore, the investigators propose to study the safety and activity of anakinra in infants and children < 2 years old with coronary artery abnormalities from KD.

ELIGIBILITY:
Inclusion Criteria:

1. Infant or child aged 1 month to 17 years, who meets clinical criteria for KD according to American Heart Association guidelines (Table 2): Fever (T≥38oC or 100.4oC) ≥ 3 days and ≥ 2 clinical criteria with left anterior descending (LAD)/right coronary artery (RCA) Z score ≥ 3.0 or an aneurysm (≥ 1.5 x the adjacent segment) of one of the coronary artery segments
2. Patient presents within the first 20 days after fever onset
3. Parent or legal guardian able and willing to provide informed consent; adolescent or child assent as appropriate
4. Post-menarchal females: Negative pregnancy test at screening and willing to use two forms of contraception during the study
5. Males engaging in sexual activity that could lead to pregnancy willing to use a condom.

Exclusion Criteria:

1. Use of an IL-1 antagonist within the 3 months prior to enrollment
2. History of chronic disease, except asthma, atopic dermatitis, autism or controlled seizure disorder
3. History of hypersensitivity to anakinra
4. History of tuberculosis (TB) or TB exposure

Ages: 1 Month to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 22 (Actual)
Dates: Start 2014-11; Primary Completion 2022-10 (Actual); Study Completion 2022-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adriana H Tremoulet, MD, Principal Investigator — UCSD; Jane C Burns, MD, Study Director — UCSD
Locations (1):
- Rady Children's Hospital San Diego, San Diego, California, United States

REFERENCES:
- [Background] Yang J, Jain S, Capparelli EV, Best BM, Son MB, Baker A, Newburger JW, Franco A, Printz BF, He F, Shimizu C, Hoshino S, Bainto E, Moreno E, Pancheri J, Burns JC, Tremoulet AH. Anakinra Treatment in Patients with Acute Kawasaki Disease with Coronary Artery Aneurysms: A Phase I/IIa Trial. J Pediatr. 2022 Apr;243:173-180.e8. doi: 10.1016/j.jpeds.2021.12.035. Epub 2021 Dec 23. PMID 34953816
- [Derived] Tremoulet AH, Jain S, Kim S, Newburger J, Arditi M, Franco A, Best B, Burns JC. Rationale and study design for a phase I/IIa trial of anakinra in children with Kawasaki disease and early coronary artery abnormalities (the ANAKID trial). Contemp Clin Trials. 2016 May;48:70-5. doi: 10.1016/j.cct.2016.04.002. Epub 2016 Apr 11. PMID 27080929

RESULTS

PARTICIPANT FLOW:
Groups:
- Dose Level 1 (Anakinra 2-4 mg/kg/Day): Participants were administered 2-4 mg/kg/day of Anakinra intravenously every 12 hours for the first 24 hours and subsequently administered subcutaneously every 24 hours.
- Dose Level 2 (Anakinra 5-7 mg/kg/Day): Participants were administered 5-7 mg/kg/day of Anakinra intravenously every 12 hours for the first 24 hours and subsequently administered subcutaneously every 24 hours.
- Dose Level 3 (Anakinra 8-11 mg/kg/Day): Participants were administered 8-11 mg/kg/day of Anakinra intravenously every 12 hours for the first 24 hours and subsequently administered subcutaneously every 24 hours.
Period: Overall Study
Arm/Group | Dose Level 1 (Anakinra 2-4 mg/kg/Day) | Dose Level 2 (Anakinra 5-7 mg/kg/Day) | Dose Level 3 (Anakinra 8-11 mg/kg/Day)
Started | 4 | 3 | 15
Completed | 4 | 3 | 15
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dose Level 1 (Anakinra 2-4 mg/kg/Day) | Dose Level 2 (Anakinra 5-7 mg/kg/Day) | Dose Level 3 (Anakinra 8-11 mg/kg/Day) | Total
Number analyzed (Participants) | 4 | 3 | 15 | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 4 | 3 | 15 | 22
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 1.5 [0.96 to 3.9] | 0.8 [0.7 to 1.6] | 1.2 [0.9 to 1.4] | 1.1 [0.9 to 1.9]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 2 | 4
  Male | 4 | 1 | 13 | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 2 | 3
  White | 2 | 1 | 7 | 10
  More than one race | 1 | 1 | 4 | 6
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 4 | 3 | 15 | 22

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Description: The primary outcome measure was the safety and tolerability of anakinra
Time Frame: within 6 weeks of treatment
Measure: Number; unit: participants
Groups:
- Dose Level 1 (Anakinra 5-7 mg/kg/Day): Participants were administered 5-7 mg/kg/day of Anakinra intravenously every 12 hours for the first 24 hours and subsequently administered subcutaneously every 24 hours.
Arm/Group | Dose Level 1 (Anakinra 2-4 mg/kg/Day) | Dose Level 1 (Anakinra 5-7 mg/kg/Day) | Dose Level 3 (Anakinra 8-11 mg/kg/Day)
Number analyzed (Participants) | 4 | 3 | 15
participants | 2 | 3 | 13

ADVERSE EVENTS:
Time Frame: 6 weeks
Description: The definition does not differ
Arm/Group | Dose Level 1 (Anakinra 2-4 mg/kg/Day) | Dose Level 2 (Anakinra 5-7 mg/kg/Day) | Dose Level 3 (Anakinra 8-11 mg/kg/Day)
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/3 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/3 | 0/15
Other Adverse Events (participants affected / at risk) | 2/4 | 3/3 | 13/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Level 1 (Anakinra 2-4 mg/kg/Day) (N=4) | Dose Level 2 (Anakinra 5-7 mg/kg/Day) (N=3) | Dose Level 3 (Anakinra 8-11 mg/kg/Day) (N=15)
Coronary artery aneurysm (Cardiac disorders) | 0 (0) | 1 (1) | 2 (2) — 3 patients had increased CAA
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 9 (9)
Emesis (Gastrointestinal disorders) | 0 (0) | 2 (2) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-09-20): https://cdn.clinicaltrials.gov/large-docs/53/NCT02179853/Prot_SAP_000.pdf